CLINICAL TRIAL: NCT00776984
Title: A Phase III Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate Efficacy and Safety of Tiotropium Inhalation Solution Delivered Via Respimat® Inhaler (5 mcg/Day) Over 48 Weeks as add-on Controller Therapy on Top of Usual Care in Patients With Severe Persistent Asthma
Brief Title: Evaluation of Tiotropium 5 µg/Day Delivered Via the Respimat® Inhaler Over 48 Weeks in Patients With Severe Persistent Asthma on Top of Usual Care (Study II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.417; 2008-001414-25 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-10-13; First posted 2008-10-22 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

ARMS (2):
- tiotropium 5mcg/day (Experimental): patient to receive double-blind treatment with either 5mcg/day tiotropium inhalation solution or placebo inhalation solution
  Interventions: Drug: tiotropium 5mcg/day
- placebo (Experimental): patient to receive double-blind treatment with either 5mcg/day tiotropium inhalation solution or placebo inhalation solution
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tiotropium 5mcg/day — Intervention = Randomisation: patient to receive double-blind treatment with either 5mcg/day tiotropium inhalation solution or placebo inhalation solution
  Arms: tiotropium 5mcg/day
Drug: placebo — Intervention = Randomisation: patient to receive double-blind treatment with either 5mcg/day tiotropium inhalation solution or placebo inhalation solution
  Arms: placebo

SUMMARY:
The trial is a randomised, double-blind, placebo-controlled, parallel-group trial to evaluate the efficacy and safety of 5 µg tiotropium over a 48-week treatment period as compared to placebo. Tiotropium inhalation solution delivered by the Respimat® inhaler will be examined as add-on controller therapy on top of usual care in patients with severe persistent asthma. The primary objective of each trial is to evaluate the long term efficacy of tiotropium over placebo on top of usual care in patients with severe persistent asthma as determined by pulmonary function testing, effects on asthma exacerbations, effects on quality of life, on asthma control and health care resource utilisation. The secondary objective of each trial is to compare the long term safety of tiotropium with placebo in this patient population.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign and date an Informed Consent Form consistent with ICH-GCP guidelines and local legislation prior to participation in the trial (i.e. prior to any trial procedures, including any pre-trial washout of medications and medication restrictions for pulmonary function test at Visit 1).
2. Male or female patients aged at least 18 years but not more than 75 years.
3. All patients must have at least a 5-year history of asthma at the time of enrolment into the trial and the diagnosis of asthma must have been made before the patient´s age of 40.
4. All patients must have a diagnosis of severe persistent asthma and must be symptomatic despite treatment with high, stable doses of inhaled corticosteroids and a long-acting beta adrenergic agent
5. All patients must have a history of one or more asthma exacerbation in the past year.
6. Patients must have evidence of treated, severe, persistent asthma in postbronchodilator pulmonary function tests.
7. Patients should be never-smokers or ex-smokers who stopped smoking at least one year prior to enrolment and who have a smoking history of less than 10 pack years
8. Patients must be able to use the Respimat® inhaler correctly
9. Patients must be able to perform all trial related procedures including technically acceptable pulmonary function tests and use of the electronic diary/peak flow meter.

Exclusion criteria:

1. Patients with a significant disease other than asthma. A significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the trial, or (ii) influence the results of the trial, or (iii) cause concern regarding the patient´s ability to participate in the trial.
2. Patients with clinically relevant abnormal screening haematology or blood chemistry.
3. Patients with a recent history (i.e. six months or less) of myocardial infarction, hospitalisation for cardiac failure during the past year, any unstable or life threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year, known active tuberculosis, malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years (treated basal cell carcinoma allowed), lung diseases other than asthma (e.g. COPD), significant alcohol or drug abuse within the past two years, patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1.
4. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the 6 weeks prior to the screening visit (Visit 1).
5. Patients using oral corticosteroid medication at stable doses exceeding 5 mg prednisolone or prednisolone equivalent every day or 10 mg prednisolone or prednisolone equivalent every second day.
6. Patients with known hypersensitivity to anticholinergic drugs, BAC, EDTA or any other components of the tiotropium inhalation solution.
7. Pregnant or nursing women or women of childbearing potential not using a highly effective method of birth control. Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation/salpingectomy, or post-menopausal for at least two years.
8. Patients who have taken an investigational drug within four weeks or six half-lives (whichever is greater) prior to Visit 1.
9. Patients who have been treated with the long-acting anticholinergic tiotropium (Spiriva®), beta-blocker medication, oral beta-adrenergics, other non-approved and according to international guidelines not recommended ´experimental´ drugs for routine asthma therapy (e.g. TNF-alpha blockers, methotrexate, cyclosporin) within four weeks prior to the Screening Visit (Visit 1) or during the screening period.
10. Patients with any asthma exacerbation or respiratory tract infection in the four weeks prior to the trial.
11. Patients who have previously been randomised in this trial or in the respective twin trial (205.416 versus 205.417) or are currently participating in another trial.
12. Patients with a known narrow-angle glaucoma.

Note:

As with other anticholinergic drugs, tiotropium should be used with caution in patients with prostatic hyperplasia or bladder neck obstruction.

As with all predominantly renally excreted drugs, patients with moderate to severe renal impairment (known creatinine clearance of <= 50 mL/min) treated with tiotropium should be monitored closely.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (75):
- United States (18):
  - 205.417.01061 Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - 205.417.01052 Boehringer Ingelheim Investigational Site, Fresno, California
  - 205.417.01051 Boehringer Ingelheim Investigational Site, Stockton, California
  - 205.417.01056 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 205.417.01065 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 205.417.01059 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 205.417.01068 Boehringer Ingelheim Investigational Site, Normal, Illinois
  - 205.417.01063 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 205.417.01064 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 205.417.01066 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 205.417.01069 Boehringer Ingelheim Investigational Site, Ocean City, New Jersey
  - 205.417.01062 Boehringer Ingelheim Investigational Site, Albany, New York
  - 205.417.01058 Boehringer Ingelheim Investigational Site, Great Neck, New York
  - 205.417.01055 Boehringer Ingelheim Investigational Site, Rockville Centre, New York
  - 205.417.01067 Boehringer Ingelheim Investigational Site, High Point, North Carolina
  - 205.417.01070 Boehringer Ingelheim Investigational Site, Canton, Ohio
  - 205.417.01053 Boehringer Ingelheim Investigational Site, Upland, Pennsylvania
  - 205.417.01054 Boehringer Ingelheim Investigational Site, Richmond, Virginia
- 205.417.61051 Boehringer Ingelheim Investigational Site, Concord, New South Wales, Australia
- Canada (3):
  - 205.417.02051 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 205.417.02053 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 205.417.02052 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- Denmark (2):
  - 205.417.45052 Boehringer Ingelheim Investigational Site, Aalborg
  - 205.417.45051 Boehringer Ingelheim Investigational Site, Aarhus C
- Germany (5):
  - 205.417.49052 Boehringer Ingelheim Investigational Site, Berlin
  - 205.417.49054 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.417.49053 Boehringer Ingelheim Investigational Site, Lübeck
  - 205.417.49051 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 205.417.49055 Boehringer Ingelheim Investigational Site, Weinheim
- Italy (4):
  - 205.417.39052 Boehringer Ingelheim Investigational Site, Bussolengo (vr)
  - 205.417.39054 Boehringer Ingelheim Investigational Site, Milan
  - 205.417.39051 Boehringer Ingelheim Investigational Site, Pavia
  - 205.417.39053 Boehringer Ingelheim Investigational Site, Pietra Ligure (sv)
- Japan (16):
  - 205.417.81063 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 205.417.81056 Boehringer Ingelheim Investigational Site, Hiroshima, Hiroshima
  - 205.417.81051 Boehringer Ingelheim Investigational Site, Itabashi-ku, Tokyo
  - 205.417.81059 Boehringer Ingelheim Investigational Site, Kagoshima, Kagoshima
  - 205.417.81053 Boehringer Ingelheim Investigational Site, Kishiwada, Osaka
  - 205.417.81057 Boehringer Ingelheim Investigational Site, Kitakyusyu, Fukuoka
  - 205.417.81058 Boehringer Ingelheim Investigational Site, Koga, Fukuoka
  - 205.417.81055 Boehringer Ingelheim Investigational Site, Kurashiki, Okayama
  - 205.417.81064 Boehringer Ingelheim Investigational Site, Kurume, Fukuoka
  - 205.417.81062 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 205.417.81052 Boehringer Ingelheim Investigational Site, Osaka-sayama, Osaka
  - 205.417.81066 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 205.417.81065 Boehringer Ingelheim Investigational Site, Seto, Aichi
  - 205.417.81060 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
  - 205.417.81061 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
  - 205.417.81054 Boehringer Ingelheim Investigational Site, Wakayama, Wakayama
- Netherlands (3):
  - 205.417.31051 Boehringer Ingelheim Investigational Site, Groningen
  - 205.417.31053 Boehringer Ingelheim Investigational Site, Leeuwarden
  - 205.417.31052 Boehringer Ingelheim Investigational Site, Schiedam
- New Zealand (4):
  - 205.417.64054 Boehringer Ingelheim Investigational Site, Auckland NZ
  - 205.417.64053 Boehringer Ingelheim Investigational Site, Christchurch
  - 205.417.64052 Boehringer Ingelheim Investigational Site, Newtown Wellington NZ
  - 205.417.64051 Boehringer Ingelheim Investigational Site, Tauranga
- Russia (3):
  - 205.417.07051 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.417.07052 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.417.07053 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Serbia (3):
  - 205.417.38153 Boehringer Ingelheim Investigational Site, Belgrade
  - 205.417.38152 Boehringer Ingelheim Investigational Site, Kamenitz
  - 205.417.38151 Boehringer Ingelheim Investigational Site, Niš
- South Africa (4):
  - 205.417.27051 Boehringer Ingelheim Investigational Site, Bellville
  - 205.417.27052 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.417.27053 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.417.27054 Boehringer Ingelheim Investigational Site, Cape Town
- Turkey (Türkiye) (3):
  - 205.417.90052 Boehringer Ingelheim Investigational Site, Ankara
  - 205.417.90053 Boehringer Ingelheim Investigational Site, Ankara
  - 205.417.90051 Boehringer Ingelheim Investigational Site, İzmit
- Ukraine (3):
  - 205.417.38053 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.417.38051 Boehringer Ingelheim Investigational Site, Kiev
  - 205.417.38052 Boehringer Ingelheim Investigational Site, Vinnytsia
- United Kingdom (3):
  - 205.417.44051 Boehringer Ingelheim Investigational Site, Chertsey
  - 205.417.44053 Boehringer Ingelheim Investigational Site, Exeter
  - 205.417.44052 Boehringer Ingelheim Investigational Site, Windsor

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Halpin DMG, Meltzer EO, Pisternick-Ruf W, Moroni-Zentgraf P, Engel M, Zaremba-Pechmann L, Casale T, FitzGerald JM. Peak expiratory flow as an endpoint for clinical trials in asthma: a comparison with FEV1. Respir Res. 2019 Jul 18;20(1):159. doi: 10.1186/s12931-019-1119-6. PMID 31319851
- [Derived] Casale TB, Bateman ED, Vandewalker M, Virchow JC, Schmidt H, Engel M, Moroni-Zentgraf P, Kerstjens HAM. Tiotropium Respimat Add-on Is Efficacious in Symptomatic Asthma, Independent of T2 Phenotype. J Allergy Clin Immunol Pract. 2018 May-Jun;6(3):923-935.e9. doi: 10.1016/j.jaip.2017.08.037. Epub 2017 Nov 22. PMID 29174062
- [Derived] Kerstjens HA, Engel M, Dahl R, Paggiaro P, Beck E, Vandewalker M, Sigmund R, Seibold W, Moroni-Zentgraf P, Bateman ED. Tiotropium in asthma poorly controlled with standard combination therapy. N Engl J Med. 2012 Sep 27;367(13):1198-207. doi: 10.1056/NEJMoa1208606. Epub 2012 Sep 2. PMID 22938706

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients treated with matching placebo
- Tio R5: Patients treated with tiotropium inhalation solution 5 microgram qd
Period: Overall Study
Arm/Group | Placebo | Tio R5
Started | 234 | 219
Completed | 203 | 198
Not Completed | 31 | 21
Not completed — Adverse Event | 8 | 2
Not completed — Protocol Violation | 4 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 12 | 7
Not completed — Lack of Efficacy | 0 | 1
Not completed — Other | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tio R5 | Total
Number analyzed (Participants) | 234 | 219 | 453
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (11.7) | 51.4 (12.5) | 52.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 127 | 262
  Male | 99 | 92 | 191

OUTCOME MEASURES:

1. Primary Outcome: Peak Forced Expiratory Volume in 1 Second (FEV1) Response Within 3 Hours Post Dosing (0-3h) After a Treatment Period of 24 Weeks.
Description: Peak FEV1 0-3h response was defined as the difference between the maximum FEV1 measured within the first 3 hours post dosing after a treatment period of 24 weeks and the FEV1 baseline measurement (10 minutes before the first dose of trial medication). Mixed Model Repeated Measure (MMRM) results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and 24 weeks
Population: All patients from Full Analysis Set (FAS) FAS is defined as all patients in the treated set who have baseline data and at least one on-treatment efficacy value.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.248 (0.024) | 0.401 (0.025)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Step-wise testing for co-primary endpoints, confirmatory only if previous hypotheses had been successful, significance level of alpha=0.05 (two-sided); Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.154, 95% CI [0.091 to 0.217], Standard Error of Mean 0.032 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

2. Primary Outcome: Trough FEV1 Response Determined After a Treatment Period of 24 Weeks.
Description: The trough FEV1 is defined as the pre-dose FEV1 measured 10 minutes before the last administration of randomised treatment. Trough FEV1 response was defined as the difference between the trough FEV1 measured after a treatment period of 24 weeks and the FEV1 baseline measurement. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and 24 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.044 (0.022) | 0.155 (0.023)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.111, 95% CI [0.053 to 0.169], Standard Error of Mean 0.030 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

3. Primary Outcome: Time to First Severe Asthma Exacerbation During the 48-week Treatment of the Pooled Data From the Two Twin Trials 205.416 (NCT00772538) and the Present 205.417 (NCT00776984).
Description: Severe asthma exacerbations were pre-defined as all asthma exacerbations that required treatment with systemic (including oral) corticosteroids for at least 3 days or (in case of ongoing and pre-existing systemic corticosteroid therapy) that required at least a doubling of the previous daily dose of systemic corticosteroids for at least 3 days.
Time Frame: 48 weeks
Population: All patients from FAS of the pooled twin studies 205.416 and 205.417. As <50percent (149 of 454 patients in the placebo group and 122 of 453 patients in the Tio R5 group) of patients had severe exacerbation, the median time was not calculable.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 454 | 453
Days | NA (NA) [NA to NA] — As <50percent (149 of 454 patients in the placebo group) of patients had severe exacerbation, the median time was not calculable. | NA (NA) [NA to NA] — As <50percent (122 of 453 patients in the Tio R5 group) of patients had severe exacerbation, the median time was not calculable.
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0343, Regression, Cox — Confirmatory only if previous hypotheses for each of the 2 twin studies had been successful, significance level of alpha=0.05 (2-sided). A pre-specified interim analysis was performed. Cui et al (Biometrics,1999) was used to calculate the p-value; Parameter estimates of Cox proportional hazard model regression regarding. Only treatment was fitted as an effect in the model; Hazard Ratio (HR) = 0.790 — If HR is below 1 then favours tiotropium

4. Secondary Outcome: Peak (Within 3 Hours Post-dosing) Forced Vital Capacity (FVC) Response at the End of the 24-week Treatment Period.
Description: Peak FVC 0-3h response was defined as the difference between the maximum FVC measured within the first 3 hours post dosing after a treatment period of 24 weeks and the FVC baseline measurement (10 minutes before the first dose of trial medication). Mixed Model Repeated Measure (MMRM) results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and 24 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.323 (0.032) | 0.416 (0.033)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0275, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.094, 95% CI [0.010 to 0.177], Standard Error of Mean 0.042 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

5. Secondary Outcome: Trough FVC Response at the End of the 24-week Treatment Period.
Description: The trough FVC is defined as the pre-dose FVC measured 10 minutes before the last administration of randomised treatment. Trough FVC response was defined as the difference between the trough FVC measured after a treatment period of 24 weeks and the FVC baseline measurement. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and 24 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.044 (0.030) | 0.150 (0.032)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0099, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.106, 95% CI [0.025 to 0.186], Standard Error of Mean 0.041 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

6. Secondary Outcome: FEV1 Area Under the Curve (AUC0-3h) Response at the End of the 24-week Treatment Period.
Description: The AUC0-3h was calculated as area under the curve from zero to 3 hours using the trapezoidal rule divided by the observation time (3 hours) to report in litres. The trough value was assigned to zero time. Response was defined as change from baseline in FEV1 AUC0-3h after a treatment period of 24 weeks. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit baseline*visit.
Time Frame: Baseline and 24 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.164 (0.022) | 0.307 (0.023)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.143, 95% CI [0.084 to 0.202], Standard Error of Mean 0.030 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

7. Secondary Outcome: FVC (AUC0-3h) Response at the End of the 24-week Treatment Period.
Description: The AUC0-3h was calculated as area under the curve from zero to 3 hours using the trapezoidal rule divided by the observation time (3 hours) to report in litres. The trough value was assigned to zero time. Response was defined as change from baseline in FVC AUC0-3h after a treatment period of 24 weeks. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit baseline*visit.
Time Frame: Baseline and 24 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.187 (0.030) | 0.295 (0.031)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0063, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.109, 95% CI [0.031 to 0.187], Standard Error of Mean 0.040 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

8. Secondary Outcome: Peak FEV1 0-3h Response at the End of the 48-week Treatment Period.
Description: Peak FEV1 0-3h response was defined as the difference between the maximum FEV1 measured within the first 3 hours post dosing after a treatment period of 48 weeks and the FEV1 baseline measurement (10 minutes before the first dose of trial medication). Mixed Model Repeated Measure (MMRM) results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and 48 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.245 (0.025) | 0.397 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.152, 95% CI [0.087 to 0.217], Standard Error of Mean 0.033 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

9. Secondary Outcome: Trough FEV1 Response at the End of the 48-week Treatment Period.
Description: The trough FEV1 is defined as the pre-dose FEV1 measured 10 minutes before the last administration of randomised treatment. Trough FEV1 response was defined as the difference between the trough FEV1 measured after a treatment period of 48 weeks and the FEV1 baseline measurement. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and 48 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.063 (0.023) | 0.155 (0.023)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.092, 95% CI [0.032 to 0.151], Standard Error of Mean 0.030 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

10. Secondary Outcome: AUC0-3h FEV1 Response at the End of the 48-week Treatment Period.
Description: The AUC0-3h was calculated as area under the curve from zero to 3 hours using the trapezoidal rule divided by the observation time (3 hours) to report in litres. The trough value was assigned to zero time. Response was defined as change from baseline in FEV1 AUC0-3h after a treatment period of 48 weeks. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit baseline*visit.
Time Frame: Baseline and 48 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.172 (0.023) | 0.310 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.138, 95% CI [0.078 to 0.199], Standard Error of Mean 0.031 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

11. Secondary Outcome: Peak FVC 0-3h Response at the End of the 48-week Treatment Period.
Description: Peak FVC 0-3h response was defined as the difference between the maximum FVC measured within the first 3 hours post dosing after a treatment period of 48 weeks and the FVC baseline measurement (10 minutes before the first dose of trial medication). MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and 48 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.305 (0.033) | 0.420 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0088, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.114, 95% CI [0.029 to 0.200], Standard Error of Mean 0.044 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

12. Secondary Outcome: Trough FVC Response at the End of the 48-week Treatment Period.
Description: The trough FVC is defined as the pre-dose FVC measured 10 minutes before the last administration of randomised treatment. Trough FVC response was defined as the difference between the trough FVC measured after a treatment period of 48 weeks and the FVC baseline measurement. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and 48 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.072 (0.031) | 0.142 (0.032)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0933, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.071, 95% CI [-0.012 to 0.153], Standard Error of Mean 0.042 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

13. Secondary Outcome: FVC AUC0-3h Response at the End of the 48-week Treatment Period.
Description: The AUC0-3h was calculated as area under the curve from zero to 3 hours using the trapezoidal rule divided by the observation time (3 hours) to report in litres. The trough value was assigned to zero time. Response was defined as change from baseline in FVC AUC0-3h after a treatment period of 48 weeks. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit baseline*visit.
Time Frame: Baseline and 48 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.190 (0.031) | 0.299 (0.032)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0074, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.109, 95% CI [0.029 to 0.189], Standard Error of Mean 0.041 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

14. Secondary Outcome: Mean Pre-dose Morning Peak Expiratory Flow (PEFa.m.) Response (Diary Data) of Last-7-days-before-week-24-visit .
Description: Weekly means obtained during the last 7 days before week 24 visit were compared (measured by patients at home using the asthma monitor device). Response was defined as change from baseline. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and last 7 days before week 24 visit
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
L/min | -3.258 (3.954) | 17.396 (4.136)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 20.654, 95% CI [11.199 to 30.108], Standard Error of Mean 4.807 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

15. Secondary Outcome: Mean Pre-dose Evening Peak Expiratory Flow (PEFp.m.) Response (Diary Data) of Last-7-days-before-week 24-visit.
Description: as for outcome 14
Time Frame: Baseline and last 7 days before week 24 visit
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
L/min | -7.295 (4.188) | 25.158 (4.397)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 32.453, 95% CI [22.532 to 42.374], Standard Error of Mean 5.044 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

16. Secondary Outcome: Mean Pre-dose FEV1 a.m. Response (Diary Data) of Last-7-days-before-week 24-visit.
Description: as for outcome 14
Time Frame: Baseline and last 7 days before week 24 visit
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | 0.006 (0.025) | 0.096 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0027, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.090, 95% CI [0.031 to 0.149], Standard Error of Mean 0.030 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

17. Secondary Outcome: Mean Pre-dose FEV1-p.m.Response (Diary Data) of Last-7-days-before-week 24-visit.
Description: as for outcome 14
Time Frame: Baseline and last 7 days before week 24 visit
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Liter | -0.015 (0.027) | 0.122 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.137, 95% CI [0.074 to 0.200], Standard Error of Mean 0.032 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

18. Secondary Outcome: Mean PEF Variability Response (Absolute Difference Between Morning and Evening PEF Value Divided by Their Mean) of Last-7-days-before-week 24-visit.
Description: Weekly means obtained during the last 7 days before week 24 visit were compared (measured by patients at home using the asthma monitor device). The PEF variability is the absolute difference between morning and evening PEF value divided by their mean, expressed as a percent. Response was defined as change from baseline. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and last 7 days before week 24 visit
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Percent | -1.808 (0.617) | -0.611 (0.641)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.1073, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 1.197, 95% CI [-0.261 to 2.655], Standard Error of Mean 0.741 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

19. Secondary Outcome: Time to First Severe Asthma Exacerbation During the 48-week Treatment.
Description: as for outcome 3
Time Frame: 48 weeks
Population: All patients from FAS. As < 50 percent (81 of 232 patients in the placebo group and 69 of 216 patients in the Tio R5 group) of patients had severe exacerbation, the median time was not calculable.
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.4788, Regression, Cox — Significance level of alpha=0.05 (two-sided); Parameter estimates of Cox proportional hazard model regarding. Only treatment was fitted as an effect in the model; Hazard Ratio (HR) = 0.89, 95% CI [0.65 to 1.23] — If HR is below 1 then favours tiotropium

20. Secondary Outcome: Number of Asthma Exacerbations Per Patient During the 48-week Treatment Period.
Description: Asthma exacerbations (including severe, non-severe; symptomatic, asymptomatic) were pre-defined as an episode of progressive increase in 1 or more asthma symptoms (e.g. shortness of breath, cough, wheezing, chest tightness or some combination of these symptoms). Additionally, decrease of patients best PEF a.m. of 30 percent or more from the patients mean PEF a.m. for at least 2 consecutive days was considered to be an objective marker of asthma exacerbation.
Time Frame: 48 weeks
Population: All patients from FAS.
Measure: Number; unit: Participants
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Participants
  0 asthma exacerbations | 82 | 106
  1 asthma exacerbation | 53 | 44
  2 asthma exacerbations | 27 | 22
  3 asthma exacerbations | 13 | 8
  4 asthma exacerbations | 14 | 10
  5 asthma exacerbations | 9 | 3
  6 asthma exacerbations | 9 | 2
  7-10 asthma exacerbations | 10 | 8
  11-20 asthma exacerbations | 13 | 11
  21+ asthma exacerbations | 2 | 2
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.1007, Poisson Regression — Significance level of alpha=0.05 (two-sided); Parameter estimates of Poisson regression model. Log exposure was used as offset and adjusted for overdispersion; Risk Ratio (RR) = 0.80, 95% CI [0.61 to 1.04], Standard Error of Mean 0.11 — Tio R5 - Placebo

21. Secondary Outcome: Number of Severe Asthma Exacerbations Per Patient During the 48-week Treatment Period.
Description: as for outcome 3
Time Frame: 48 weeks
Population: All patients from FAS.
Measure: Number; unit: Participants
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Participants
  0 severe asthma exacerbations | 151 | 147
  1 severe asthma exacerbation | 51 | 38
  2 severe asthmaexacerbations | 19 | 17
  3 severe asthma exacerbations | 5 | 8
  4 severe asthma exacerbations | 3 | 3
  5 severe asthma exacerbations | 2 | 1
  6 severe asthma exacerbations | 0 | 1
  7-10 severe asthma exacerbations | 0 | 1
  11-20 severe asthma exacerbations | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.7906, Poisson Regression — Significance level of alpha=0.05 (two-sided); Parameter estimates of Poisson regression model. Log exposure was used as offset and adjusted for overdispersion; Risk Ratio (RR) = 0.96, 95% CI [0.71 to 1.30], Standard Error of Mean 0.15 — Tio R5 - Placebo

22. Secondary Outcome: Number of Patients With at Least One Asthma Exacerbation During the 48-week Treatment Period.
Description: as for outcome 20
Time Frame: 48 weeks
Population: All patients from FAS.
Measure: Number; unit: Participants
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Participants | 150 | 110
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0040, Fisher Exact — Significance level of alpha=0.05 (two-sided); Exact 95 percent confidence interval by Clopper and Pearson; Odds Ratio (OR) = 0.57, 95% CI [0.38 to 0.84] — Tio R5 vs Placebo

23. Secondary Outcome: Number of Patients With at Least One Severe Asthma Exacerbation During the 48-week Treatment Period.
Description: as for outcome 3
Time Frame: 48 weeks
Population: All patients from FAS.
Measure: Number; unit: Participants
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Participants | 81 | 69
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.5481, Fisher Exact — Significance level of alpha=0.05 (two-sided); Exact 95 percent confidence interval by Clopper and Pearson; Odds Ratio (OR) = 0.88, 95% CI [0.58 to 1.32] — Tio R5 vs Placebo

24. Secondary Outcome: Time to First Hospitalisation for Asthma Exacerbation During the 48-week Treatment Period.
Description: as for outcome 20
Time Frame: 48 weeks
Population: All patients from FAS. As < 50 percent (10 of 232 patients in the placebo group and 8 of 216 patients in the Tio R5 group) of patients had severe exacerbation, the median time was not calculable.
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.7188, Regression, Cox — Significance level of alpha=0.05 (two-sided); Parameter estimates of Cox proportional hazard model regarding. Only treatment was fitted as an effect in the model; Hazard Ratio (HR) = 0.84, 95% CI [0.33 to 2.14] — If HR is below 1 then favours tiotropium

25. Secondary Outcome: Number of Hospitalisations for Asthma Exacerbations Per Patient During the 48-week Treatment Period.
Time Frame: 48 weeks
Population: All patients from FAS.
Measure: Number; unit: Participants
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Participants
  0 hospitalisations | 222 | 208
  1 hospitalisations | 9 | 6
  2+ hospitalisations | 1 | 2
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.8503, Poisson Regression — Significance level of alpha=0.05 (two-sided); Parameter estimates of Poisson regression model. Log exposure was used as offset and adjusted for overdispersion; Risk Ratio (RR) = 0.95, 95% CI [0.59 to 1.54], Standard Error of Mean 0.23 — Tio R5 - Placebo

26. Secondary Outcome: Number of Patients With at Least One Hospitalisation for Asthma Exacerbation During the 48-week Treatment Period.
Time Frame: 48 weeks
Population: All patients from FAS.
Measure: Number; unit: Participants
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Participants | 10 | 8
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.8129, Fisher Exact — Significance level of alpha=0.05 (two-sided); Exact 95 percent confidence interval by Clopper and Pearson; Odds Ratio (OR) = 0.85, 95% CI [0.29 to 2.46] — Tio R5 vs Placebo

27. Secondary Outcome: Quality of Life as Assessed by Standardised Asthma Quality of Life Questionnaire (AQLQ(S)) at the End of the 24-week Treatment Period.
Description: The AQLQ(S) total score was calculated as the mean of the responses to 32 questions for the domains Symptoms, Activity Limitations, Emotional Function and Environmental Stimuli and was analysed as an absolute value. The AQLQ(S) total score ranges from 1 (worst controlled) to 7 (best). MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: 24 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Scores on a scale | 4.869 (0.058) | 5.047 (0.061)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0225, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.178, 95% CI [0.025 to 0.331], Standard Error of Mean 0.078 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

28. Secondary Outcome: AQLQ(S) Total Score at the End of the 48-week Treatment Period.
Description: as for outcome 27
Time Frame: 48 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Scores on a scale | 4.945 (0.060) | 5.085 (0.062)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0803, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.140, 95% CI [-0.017 to 0.296], Standard Error of Mean 0.080 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

29. Secondary Outcome: Asthma Control as Assessed by Asthma Control Questionnaire (ACQ) at the End of the 24-week Treatment Period.
Description: For the ACQ, the total score was calculated as the mean of the responses to 7 questions and was analysed as an absolute value. The score ranges from 0 (no impairment) to 6 (maximum impairment). MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: 24 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Score on a scale | 2.210 (0.050) | 2.011 (0.052)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0030, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = -0.199, 95% CI [-0.330 to -0.068], Standard Error of Mean 0.067 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

30. Secondary Outcome: ACQ Score at the End of the 48-week Treatment Period.
Description: as for outcome 29
Time Frame: 48 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Scores on a scale | 2.159 (0.051) | 2.027 (0.053)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0533, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = -0.133, 95% CI [-0.267 to 0.002], Standard Error of Mean 0.069 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

31. Secondary Outcome: Asthma Symptom Free Days Response During the Last-7-days-before-week-24-visit .
Description: Weekly means obtained during the last 7 days before week 24 visit were compared (measured by patients at home using the asthma monitor device). The response is defined as the change of the weekly mean from the baseline weekly mean. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and last 7 days before week 24 visit
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Days | 0.065 (0.023) | 0.077 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.6632, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.012, 95% CI [-0.043 to 0.067], Standard Error of Mean 0.028 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

32. Secondary Outcome: Mean Pro Re Nata (as Needed, PRN) Rescue Medication Use Response During the Last-7-days-before-week-24-visit .
Description: Weekly means obtained during the last 7 days before week 24 visit were compared. The response is defined as the change of the weekly mean from the baseline weekly mean. The use of PRN salbutamol (albuterol rescue medication) is determined by the number of puffs of rescue therapy used per day. MMRM results. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and last 7 days before week 24 visit
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: Puffs
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 232 | 216
Puffs | -0.881 (0.158) | -1.144 (0.163)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.1664, Mixed Models Analysis — Significance level of alpha=0.05 (two-sided); REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = -0.263, 95% CI [-0.635 to 0.110], Standard Error of Mean 0.189 — Tio R5 - Placebo. Means are adjusted for treatment, centre, visit, baseline, treatment*visit and baseline*visit

33. Post Hoc Outcome: The Responder Rate as Assessed by the ACQ From the Two Twin Trials 205.416 (NCT00772538) and the Present 205.417 (NCT00776984)
Description: The responder rate as assessed by the Asthma Control Questionnaire (ACQ) determined at 24-weeks and 48-weeks (on combined data from the two twin trials 205.416 (NCT00772538) and 205.417 (NCT00776984)). A patient was considered to be a responder if he or she was reported with an improvement (decrease) in the ACQ total score of at least 0.5 points.
  The ACQ total score was calculated as the mean of the responses to 7 questions and was analysed as an absolute value. The score ranges from 0 (no impairment) to 6 (maximum impairment).
  This outcome definition is taken from the primary outcome definition for the twin trials 205.418 (NCT01172808) and 205.419 (NCT01172821) of the same development program.
Time Frame: 24 weeks, 48 weeks
Population: FAS of combined data from the two twin trials 205.416 (NCT00772538) and 205.417 (NCT00776984)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tio R5
Number analyzed (Participants) | 454 | 453
percentage of participants
  24 weeks | 46.9 | 53.9
  48 weeks | 45.2 | 58.1
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Comparison at 24 weeks; Test type: Superiority or Other; p = 0.0427, Fisher Exact — Calculated as 2*one-sided-p-value in the direction corresponding to testing the null hypothesis; Odds Ratio (OR) = 1.32, 95% CI 2-sided [1.01 to 1.73] — Tio R5 / Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; Comparison at 48 weeks; Test type: Superiority or Other; p = 0.0001, Fisher Exact — Calculated as 2*one-sided-p-value in the direction corresponding to testing the null hypothesis; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.28 to 2.21] — Tio R5 / Placebo

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Placebo | Tio R5
Serious Adverse Events (participants affected / at risk) | 25/234 | 19/219
Other Adverse Events (participants affected / at risk) | 171/234 | 134/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=234) | Tio R5 (N=219)
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Abscess limb (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Labile hypertension (Vascular disorders) | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=234) | Tio R5 (N=219)
Bronchitis (Infections and infestations) | 10 | 13
Nasopharyngitis (Infections and infestations) | 36 | 32
Sinusitis (Infections and infestations) | 12 | 13
Peak expiratory flow rate decreased (Investigations) | 64 | 44
Headache (Nervous system disorders) | 20 | 17
Asthma (Respiratory, thoracic and mediastinal disorders) | 112 | 83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.